CLINICAL TRIAL: NCT00117234
Title: A Study to Assess the Impact of Subcutaneous (SC) Darbepoetin Alfa Treatment on Exercise Tolerance and Left Ventricular Structure in Subjects With Symptomatic Congestive Heart Failure (CHF) and Anemia
Brief Title: Impact of Darbepoetin Alfa on Exercise Tolerance and Left Ventricular Structure in Subjects With Symptomatic Congestive Heart Failure (CHF) and Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020126
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Congestive Heart Failure; Anemia
Keywords: chronic heart failure; congestive heart failure; low hemoglobin; anemia; CHF; Symptomatic Congestive Heart Failure (CHF)
MeSH Terms: conditions — Heart Failure; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
The purpose of this study was to evaluate the effect of treatment with darbepoetin alfa on peak oxygen consumption (peak VO2) in subjects with symptomatic CHF and anemia.

ELIGIBILITY:
Inclusion Criteria: - Symptomatic CHF for at least 3 months - Reduced left ventricular ejection fraction - Stable heart failure medication - Peak VO2 less than or equal to 16 ml/kg/min - Hemoglobin concentration between 9.0 and 12.0 g/dL Exclusion Criteria: - Hypertension - Unstable angina pectoris or recent myocardial infarction - Likely to receive cardiac transplant - Unable to do cardiopulmonary exercise testing - Major organ transplant (e.g., lung, liver, heart) or renal replacement therapy (e.g., dialysis) - Recent or current treatment for malignancy - Systemic hematologic disease - Anemia due to acute or chronic bleeding - Recent Epogen® or darbepoetin alfa therapy - Recent blood transfusion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Study Completion 2004-07

PRIMARY OUTCOMES:
Exercise tolerance, measured as peak VO(subscript)2

SECONDARY OUTCOMES:
Exercise duration; *NYHA classification; *Patient-reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Ponikowski P, Anker SD, Szachniewicz J, Okonko D, Ledwidge M, Zymlinski R, Ryan E, Wasserman SM, Baker N, Rosser D, Rosen SD, Poole-Wilson PA, Banasiak W, Coats AJ, McDonald K. Effect of darbepoetin alfa on exercise tolerance in anemic patients with symptomatic chronic heart failure: a randomized, double-blind, placebo-controlled trial. J Am Coll Cardiol. 2007 Feb 20;49(7):753-62. doi: 10.1016/j.jacc.2006.11.024. Epub 2007 Feb 5. PMID 17306703
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20020126.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf